CLINICAL TRIAL: NCT03707535
Title: A Randomized, Controlled, Double-Blind, Phase 3 Study to Compare the Efficacy, Pharmacokinetics and Safety Between CT-P13 and China Approved Remicade When Co-administered With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: To Compare the Efficacy, Pharmacokinetics and Safety Between CT-P13 and China Approved Remicade When Co-administered With Methotrexate in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P13 3.6
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CT-P13; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P13 (Experimental)
  Interventions: Biological: CT-P13
- China-approved Remicade (Active Comparator)
  Interventions: Biological: Remicade

INTERVENTIONS:
Biological: CT-P13 — 3 mg/kg, 2-hour infusion per dose co-administered with methotrexate and folic acid
  Arms: CT-P13
Biological: Remicade — 3 mg/kg, 2-hour infusion per dose co-administered with methotrexate and folic acid
  Arms: China-approved Remicade

SUMMARY:
To demonstrate that CT-P13 is equivalent to China-approved Remicade at Week 14, in terms of efficacy as determined by clinical response according to the change from baseline in disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of rheumatoid arthritis
* Has active disease as defined in DAS28 Criteria

Exclusion Criteria:

* Has a history of tuberculosis (TB) or a current diagnosis of TB
* Has previously received a biological agent
* Has previously received a tumor necrosis factor alpha (TNF α) inhibitor
* Allergies to any of the excipients of infliximab or hypersensitivity to murine and/or human proteins or immunoglobulin products
* Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment: DAS28 (CRP) at Week 14 | Week 14
  Clinical response according to the change from baseline in disease activity as measured by the Disease Activity Score using 28 joint counts (DAS28) (C-reactive protein[CRP])

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No